CLINICAL TRIAL: NCT04357054
Title: Darwish Hysteroscopic Test (Hysteroscopic Bubble Suction and Tubal Peristalsis of Darwish Triad) in Myomatous Uterus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Darwish test in myoma
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Tubal Patency and Peristalsis During Hysteroscopy
Keywords: hysteroscopy; tubal patency; bubble suction test; tubal peristalsis; liomyoma; Darwish test

STUDY DESIGN:
Intervention Model Description: hysteroscopic bubble suction and tubal peristalsis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal uterus (Active Comparator): Darwish test
  Interventions: Diagnostic Test: Darwish test
- Myomatous uterus (Active Comparator): Darwish test
  Interventions: Diagnostic Test: Darwish test

INTERVENTIONS:
Diagnostic Test: Darwish test — Infertile women planned for combined laparoscopy and hysteroscopy as an integral part of infertility wok-up.
  Other Names: hysteroscopic bubble suction and tubal peristalsis of Darwish triad

SUMMARY:
This study aims to test the impact of different types of liomyoma on Darwish test (hysteroscopic bubble suction test and tubal peristalsis of Darwish triad ) in women subjected to postmenstrual combined laparoscopy and hysteroscopy.

DETAILED DESCRIPTION:
It will include infertile women planned for combined laparoscopy and hysteroscopy as an integral part of infertility wok-up. Preoperative counseling of all patients followed by an informed written consent taken from those who will agree. The included patients subjected to complete history taking and meticulous physical examination. A suspected pregnancy, active pelvic inflammatory disease (PID), severe co-morbidity, e.g., severe cardiac, neurologic, or chest disease, and other medical contraindications to pregnancy will be exclusion criteria of this study. All cases should have basic TVS examination, normal husband's semen analysis, and a recent HSG. Basic TVs should comment on any uterine pathology . If a uterine myoma is seen with its characteristic hypoechoic, but can be isoechoic, or even hyperechoic shadow compared to normal myometrium. Calcification is seen as echogenic foci with posterior shadowing. Cystic areas of necrosis or degeneration may be seen. Definition of the number, site and proximity to corneal ends of the uterus should be addressed.

Sample size calculation based on our previous study on the prevalence of tubal patency using bubble suction test in infertility patients with normal FT (5). The percentage of agreement between office hysteroscopy and diagnostic laparoscopy will be 92% and 88% for the right and left tubes respectively. If it is supposed that bubble suction test would be positive in about 90% of apparently normal FT and it would be positive in about 60% of cases with liomyomata, sample size in each group would be 51 cases needed to have a confidence level of 95% with α error of 0.05 (the real value is within ±5% of the measured/surveyed value). Eligible women will subjected to combined laparoscopy and hysteroscopy essentially postmenstrual. Since this study will include infertility patients consenting for all options of endoscopic management of any infertility problem, a decision of general anesthesia will be made in all cases. The abdomen, vulva, vagina and the thighs will be disinfected with a 10% povidone-iodine solution. Sterile draping will be applied. The procedure started by a standard double puncture laparoscopy to search for any possible cause of infertility. An additional auxiliary portal will be made whenever a therapeutic procedure is needed. After completion of laparoscopic procedures to enhance fertility like myomectomy, adhesiolysis or management of endometriosis, tubal perchromation test using methylene blue dye will be done with comment on tubal patency in both sides. FT length, integrity, size, external surface and fimbriae will be reported bilaterally.

Thereafter, conventional diagnostic hysteroscopy will be performed using a 4mm 30° rigid scope with a 5mm outer sheath (Karl Storz, Tutlingen, Germany), and the uterus will be distended with normal saline at 100-150 mmHg generated from a pneumatic cuff of sphygmomanometer wrapped around the 500-cm3 infusion bottle. As attached to a 250-W Xenon light source, the scope will be introduced gently through the cervical canal and internal os as previously described (5). To perfectly perform hysteroscopic tubal patency testing the following tricks should be followed. Clear view of the endometrial cavity should be achieved on panoramic view by placing the hysteroscope at internal os waiting for a while to achieve homogenous distension. The uterine cavity should be systematically examined starting by its anterior and posterior walls, the fundus, and the borders. Examination will be considered complete if the both tubal ostia will be reached describing any gross pathology, e.g., septum, adhesions, polyp, myoma, and growth.

If the uterus appears externally and internally normal , the patient allocated as group A. If there is one or more liomyomata the patient allocated as group B.

Prerequisites for a successful access to evaluate tubal patency include utilization of a 300 telescope with gaining skill of its rotation to reach both cornea and most importantly orientation with a fundamental anatomic triad (Darwish triad) (DT). The most proximal corneal fine wide circle is the ostium (the end of the endometrial cavity) representing a base of a cone which is followed by a shallow conical groove (the first millimeters of the intramural part of FT). Finally, a distal pinhole dark spot (the narrowest part of the FT) representing the tip of the cone. Putting DT (ostium, intramural part and dark spot) in mind is the key step to evaluate tubal patency and physiology via hysteroscopy. If DT is clearly accessible, the hysteroscopist should comment on this. If there are some osteal lesions like tiny polypi or fine adhesions (figure 3, video 2) that may hinder proper evaluation of the tubal anatomy and physiology, the hysteroscopist should notice and document. Passage of any air bubbles in the irrigating fluid towards DT is reported. If no observed air bubbles, the hysteroscopist should inject just 2 ml of air into the rubber end of the sterile infusion set. Hysteroscopic bubble suction test is considered positive if air bubbles are sucked by DT within 1 min. During this period, neither injection of air nor increased pressure will be done. If no suction of gas bubbles occurred, the examiner should wait for 1 min more to exclude tubal spasm. Again, if no suction of the bubbles by DT and their accumulation at the corneal end, the test will be considered negative (figure 4). Simultaneously, careful visualization of any change in the shape of the ostium and intramural part of FT particularly during suction of the air bubbles will be recorded in all cases. Tubal peristalsis is defined as observed osteal and intramural tubal rhythmic opening and closing on maintained intrauterine pressure, i.e., periodic changes of DT in the form of widening followed by collapse on meticulous observation. If the ostium and intramural part of the tube is obviously opened followed by collapse and non-visualization of the pinhole dark spot of DT for a while, positive peristalsis will be reported. The same steps repeated on the contralateral side and reported.

ELIGIBILITY:
Inclusion Criteria:

* infertile women planned for combined laparoscopy and hysteroscopy as an integral part of infertility wok-up.

Exclusion Criteria:

* A suspected pregnancy, active pelvic inflammatory disease (PID), severe co-morbidity, e.g., severe cardiac, neurologic, or chest disease, and other medical contraindications to pregnancy will be exclusion criteria of this study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-05 (Estimated); Primary Completion 2023-05-23 (Estimated); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
positive bubble suction and tubal peristalsis (Darwish test) in women with myomata and those without. | 1 month
  Diagnostic tubal patency test via hysteroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No